CLINICAL TRIAL: NCT01748292
Title: A Phase IIIb, Multicenter, Randomized, Controlled Study of the Safety, Tolerability and Efficacy of IVT 0.5mg Ranibizumab Monthly Compared to a Treat & Extend Protocol in Patients With Wet Age-related Macular Degeneration (T-REX)
Brief Title: Treat & Extend Treatment With 0.5mg Ranibizumab vs Monthly Treatment With 0.5mg Ranibizumab
Acronym: T-REX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Charles C Wykoff, PhD, MD (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Charles C Wykoff, PhD, MD, Deputy Director of Research, Greater Houston Retina Research
Organization: Greater Houston Retina Research (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML28513
Record Dates: First submitted 2012-12-07; First posted 2012-12-12 (Estimated); Results first posted 2017-10-20 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: Macular Degeneration
Keywords: Age related; Macular; sub retinal fluid; Age related Macular degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Monthly IVT ranibizumab (Active Comparator): Monthly intravitreal injections (IVT) ranibizumab for 24 months, not less than 21 days apart to not more than 35 days apart
  Interventions: Drug: 0.5 mg ranibizumab
- Treat and Extend IVT ranibizumab (Experimental): 0.5 mg intravitreal injections (IVT) ranibizumab for 3 consecutive months followed by a treat and extend protocol in which follow-up intervals are increased when there is no clinical and SD-OCT evidence of disease activity by 2-week intervals and patients are treated at every visit. (Comparator arm)
  Interventions: Drug: 0.5 mg ranibizumab

INTERVENTIONS:
Drug: 0.5 mg ranibizumab — Subject will receive drug (ranibizumab) via intravitreal injections (IVT) at every visit.
  Other Names: Lucentis

SUMMARY:
TREX is a phase IIIb, multicenter, randomized, controlled clinical study. Subjects will be randomized 1:2 to "monthly" (control arm) or "treat and extend" protocol (comparator arm) respectively. TREX assess the safety, tolerability and efficacy of intravitreal injections (IVT) of 0.5mg ranibizumab given monthly for up to 100 weeks followed by pro re nata (PRN) treatment for 56 weeks compared to a Treat and Extend protocol for 156 weeks in patients with wet age-related macular degeneration (AMD). Subjects treated in a treat and extend protocol receive 3 consecutive IVT 0.5 mg ranibizumab (visits 2, 4 and 5). Starting at week 8, if a subject has achieved a "dry" macula; signs of active exudation have resolved will begin a Treat and Extend protocol (visits lengthened by 2 week intervals every visit a dry macular is maintained). At the beginning of the 104-week endpoint subjects initially randomized to the TREX cohort will transition to PRN re-treatment when there is no exudative disease activity at the 12-week interval.

DETAILED DESCRIPTION:
This trial will compare the results of 2 cohorts, with different treatment intervals, to assess the safety, tolerability and efficacy of IVT of ranibizumab for the treatment of wet AMD. Specifically, this trial will evaluate the ability to reduce the amount of visits and IVT ranibizumab treatments needed all while maintaining an exudation-free macula. Subjects in both cohorts will be followed for a total of 156 weeks.

Cohort A (control arm, monthly, n=20) Subjects will receive monthly treatment of IVT 0.5 mg ranibizumab from Day 0 to week 100. Monthly treatment is defined as every 28 days (±7 days). Dosing should not occur earlier than 21 days after the previous treatment.

Week 104 - Week 156 Starting at week 104 subjects will be seen monthly and treated with IVT ranibizumab pro re nata (PRN) based on pre-defined re-treatment criteria.

Retreatment criteria for PRN phase

Re-treatment will be initiated if any of the following criteria are meet:

* Presence of any abnormal intraretinal or subretinal fluid on high resolution SD-OCT.
* Presence of new intraretinal or subretinal hemorrhage related to AMD on examination.
* 10 letter loss from previous visit, related to active wet AMD in the opinion of the treating investigator

Cohort B (comparator arm, TREX, n=40) Subjects will receive a minimum of 3 consecutive IVT 0.5 mg ranibizumab (visits 2, 4 and 5). Starting at week 8, if a subject has achieved a "dry" macula; signs of active exudation have resolved by both ophthalmic exam and SD-OCT evaluation they will begin a Treat and Extend protocol.

For a macula to be considered "dry" it must meet both the following criteria:

1. Resolution of intraretinal and subretinal fluid
2. Resolution of all subretinal hemorrhage related to active exudative AMD

Resolution of pigment epithelial detachments (PED) is not required for a macula to be considered "dry". Small intraretinal cystic areas observed on SD-OCT are acceptable and the corresponding macula can be considered dry. The criteria for these are specific; see reference images (Appendix D) for examples of acceptable intraretinal cystic spaces. When cysts described in Appendix D are present the macula should be considered dry and should be notated on the SD-OCT interpretation. Also, minimal increased retinal thickening on SD-OCT without definitive intraretinal or subretinal exudative fluid can be observed and the corresponding macula will be considered dry.

Once a "dry" macula is achieved the interval between visits is then lengthened by 2-week increments, at every visit the macula is "dry". IVT ranibizumab will be rendered at every visit, no earlier than 7 days before the target date and no later than 7 days after the target date; the interval between visits is individualized based on each patient's response to treatment. The interval between injections will not exceed 12 weeks

After a subject is extended beyond 4-weeks and develops recurrent exudative disease activity, the eye is treated and the treatment interval for the next visit is reduced by 2 weeks, compared to the previous treatment interval. The interval between treatments will be reduced by 2-week intervals until a dry macula is again established. Once a dry macula is again achieved, the interval between visits will be extended by 1-week intervals, instead of 2-week intervals.

For example: If recurrent exudative disease activity is detected after an 8-week interval, the eye is treated and the interval for the next visit is reduced to 6 weeks; if the macula is then dry after the 6-week interval, the interval is increased to 7 weeks. If the macula is then dry after the 7-week interval, the interval is increased to 8 weeks, etc.

Once an eye is extended by 1-week intervals, if recurrent exudative disease is detected again, the treatment interval for the next visit is reduced by 1 week, compared to the previous treatment interval, and will continue to be decreased by 1-week intervals until dry or the 4-week interval is reached. Once a dry macula is again established, the most recent interval between treatments is maintained for one additional visit; if the macula remains dry at this time, the interval will then be extended by 1-week increments.

If an eye exhibits recurrent exudative disease activity 3 times at a given interval and is unable to extend beyond that interval, the eye will continue treatment at the next shorter interval for 3 consecutive visits. After these 3 visits, the interval between visits will again be extended by 1-week intervals, while the macula remains "dry". If the eye exhibits recurrent exudative disease activity, the interval will be decreased by 1-week intervals until the macula is again "dry." The eye will then continue treatment at this interval for 3 consecutive visits before extending by 1-week again. This pattern of repeating 3 visits at the same "dry" interval will be repeated each time after the eye becomes "wet" before again attempting another 1-week extension.

Evidence of recurrent exudative activity

Clinical evidence of recurrent exudative disease activity requiring reducing the interval between treatments includes any of the following:

1. Evidence of subretinal or intraretinal fluid on SD-OCT which is not classified as small intraretinal cystic areas unrelated to active exudative AMD (Appendix D) or minimal increased retinal thickening by SD-OCT without definitive intraretinal or subretinal fluid
2. New macular hemorrhage related to active exudative AMD.
3. ETDRS VA loss of 5 letters from the previous measurement due to neovascular AMD disease process with corresponding SD-OCT evidence of fluid in the macula.
4. Increase in CRT of 50 microns due to active exudative AMD.

The isolated presence of a PED, or enlargement of a PED, does not constitute evidence of exudative disease activity.

If an eye has an ETDRS VA decrease of ≥ 4 lines (20 letters) or a subretinal macular hemorrhage of 1DD or larger, at any point during the trial, the subject will subsequently be treated with ranibizumab every 4 weeks.

Week 104 - Week 156 Starting at Week 104 subjects who have achieved a "dry" macula, at the 12 week interval will be seen monthly and treated pro re nata (PRN) based on pre-defined re-treatment criteria. Study visits should be scheduled to occur every 28 (±7) days relative to the date of week 104 visit.

Retreatment criteria for PRN phase

Re-treatment will be initiated if any of the following criteria are met:

* Presence of any abnormal intraretinal or subretinal fluid on high resolution SD- OCT.
* Presence of new intraretinal or subretinal hemorrhage related to AMD on examination.
* 10 letter loss from previous visit, related to active wet AMD in the opinion of the treating investigator

Starting at Week 104, subjects who have NOT achieved extension to the 12-week treatment interval will continue with the treat and extend protocol. At any time during weeks 104 to 156 if a subject achieves a "dry" macula, at the 12-week interval, they will immediately begin monthly PRN treatment based on pre-defined re-treatment criteria. Study visits should be scheduled to occur every 28 (±7) days, relative to the date the 12-week interval is achieved. Subjects will not be treated at the visit they achieve the 12 week interval (this is the date PRN treatment will begin).

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age > 50 years
* Ability and willingness to return for all scheduled visits and assessments
* Any CNVM lesion (Occult, Minimally Classic or Classic) (i.e., leakage on fluorescein angiography or subretinal, intraretinal activity on SDOCT) secondary to age-related macular degeneration.

Best corrected visual acuity in the study eye, using ETDRS testing, between 20/32 and 20/400 (Snellen equivalent), inclusive.

-The total area of subretinal hemorrhage and fibrosis must comprise less than 50% of the total lesion. Clear ocular media and adequate pupillary dilation to permit good quality fundus imaging.

Exclusion Criteria:

* Subretinal hemorrhage in the study eye that involves the center of the fovea, if the size of the hemorrhage is either > 50% of the total area of the lesion or > 1 disc area (2.54 mm2) in size
* Subfoveal fibrosis or atrophy in the study eye
* CNV in either eye due to other causes, such as ocular histoplasmosis, trauma, or pathologic myopia

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles C Wykoff, PhD, MD, Principal Investigator — Retinal Consultants of Houston
Locations (4):
- United States (4):
  - Palmetto Retina Center, West Columbia, South Carolina
  - Retina Consultants of Houston/The Medical Center, Houston, Texas
  - Retina Consultants of Houston/Katy office, Katy, Texas
  - Retina Consultants of Houston, The Woodlands, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brown DM, Kaiser PK, Michels M, Soubrane G, Heier JS, Kim RY, Sy JP, Schneider S; ANCHOR Study Group. Ranibizumab versus verteporfin for neovascular age-related macular degeneration. N Engl J Med. 2006 Oct 5;355(14):1432-44. doi: 10.1056/NEJMoa062655. PMID 17021319
- [Background] Rosenfeld PJ, Brown DM, Heier JS, Boyer DS, Kaiser PK, Chung CY, Kim RY; MARINA Study Group. Ranibizumab for neovascular age-related macular degeneration. N Engl J Med. 2006 Oct 5;355(14):1419-31. doi: 10.1056/NEJMoa054481. PMID 17021318
- [Background] Boyer DS, Heier JS, Brown DM, Francom SF, Ianchulev T, Rubio RG. A Phase IIIb study to evaluate the safety of ranibizumab in subjects with neovascular age-related macular degeneration. Ophthalmology. 2009 Sep;116(9):1731-9. doi: 10.1016/j.ophtha.2009.05.024. Epub 2009 Jul 29. PMID 19643495
- [Background] Regillo CD, Brown DM, Abraham P, Yue H, Ianchulev T, Schneider S, Shams N. Randomized, double-masked, sham-controlled trial of ranibizumab for neovascular age-related macular degeneration: PIER Study year 1. Am J Ophthalmol. 2008 Feb;145(2):239-248. doi: 10.1016/j.ajo.2007.10.004. PMID 18222192
- [Background] Schmidt-Erfurth U, Eldem B, Guymer R, Korobelnik JF, Schlingemann RO, Axer-Siegel R, Wiedemann P, Simader C, Gekkieva M, Weichselberger A; EXCITE Study Group. Efficacy and safety of monthly versus quarterly ranibizumab treatment in neovascular age-related macular degeneration: the EXCITE study. Ophthalmology. 2011 May;118(5):831-9. doi: 10.1016/j.ophtha.2010.09.004. Epub 2010 Dec 13. PMID 21146229
- [Background] Busbee BG, Yee W, Li Z, et al. Efficacy and safety of 2.0mg or 0.5mg ranibizumab in patients with subfoveal neovascular AMD: HARBOR Study. American Academy of Ophthalmology; Orlando, Florida October 24, 2011.
- [Background] Lalwani GA, Rosenfeld PJ, Fung AE, Dubovy SR, Michels S, Feuer W, Davis JL, Flynn HW Jr, Esquiabro M. A variable-dosing regimen with intravitreal ranibizumab for neovascular age-related macular degeneration: year 2 of the PrONTO Study. Am J Ophthalmol. 2009 Jul;148(1):43-58.e1. doi: 10.1016/j.ajo.2009.01.024. Epub 2009 Apr 18. PMID 19376495
- [Background] CATT Research Group; Martin DF, Maguire MG, Ying GS, Grunwald JE, Fine SL, Jaffe GJ. Ranibizumab and bevacizumab for neovascular age-related macular degeneration. N Engl J Med. 2011 May 19;364(20):1897-908. doi: 10.1056/NEJMoa1102673. Epub 2011 Apr 28. PMID 21526923
- [Background] Comparison of Age-related Macular Degeneration Treatments Trials (CATT) Research Group; Martin DF, Maguire MG, Fine SL, Ying GS, Jaffe GJ, Grunwald JE, Toth C, Redford M, Ferris FL 3rd. Ranibizumab and bevacizumab for treatment of neovascular age-related macular degeneration: two-year results. Ophthalmology. 2012 Jul;119(7):1388-98. doi: 10.1016/j.ophtha.2012.03.053. Epub 2012 May 1. PMID 22555112
- [Background] Aiello LP, Avery RL, Arrigg PG, Keyt BA, Jampel HD, Shah ST, Pasquale LR, Thieme H, Iwamoto MA, Park JE, et al. Vascular endothelial growth factor in ocular fluid of patients with diabetic retinopathy and other retinal disorders. N Engl J Med. 1994 Dec 1;331(22):1480-7. doi: 10.1056/NEJM199412013312203. PMID 7526212
- [Background] Spaide R. Ranibizumab according to need: a treatment for age-related macular degeneration. Am J Ophthalmol. 2007 Apr;143(4):679-80. doi: 10.1016/j.ajo.2007.02.024. No abstract available. PMID 17386275
- [Background] Engelbert M, Zweifel SA, Freund KB. "Treat and extend" dosing of intravitreal antivascular endothelial growth factor therapy for type 3 neovascularization/retinal angiomatous proliferation. Retina. 2009 Nov-Dec;29(10):1424-31. doi: 10.1097/IAE.0b013e3181bfbd46. PMID 19898180
- [Background] Oubraham H, Cohen SY, Samimi S, Marotte D, Bouzaher I, Bonicel P, Fajnkuchen F, Tadayoni R. Inject and extend dosing versus dosing as needed: a comparative retrospective study of ranibizumab in exudative age-related macular degeneration. Retina. 2011 Jan;31(1):26-30. doi: 10.1097/IAE.0b013e3181de5609. PMID 20890246
- [Background] Gupta OP, Shienbaum G, Patel AH, Fecarotta C, Kaiser RS, Regillo CD. A treat and extend regimen using ranibizumab for neovascular age-related macular degeneration clinical and economic impact. Ophthalmology. 2010 Nov;117(11):2134-40. doi: 10.1016/j.ophtha.2010.02.032. Epub 2010 Jul 1. PMID 20591490
- [Background] Shienbaum G, Gupta OP, Fecarotta C, Patel AH, Kaiser RS, Regillo CD. Bevacizumab for neovascular age-related macular degeneration using a treat-and-extend regimen: clinical and economic impact. Am J Ophthalmol. 2012 Mar;153(3):468-473.e1. doi: 10.1016/j.ajo.2011.08.011. Epub 2011 Oct 11. PMID 21996309
- [Derived] Wykoff CC, Ou WC, Croft DE, Payne JF, Brown DM, Clark WL, Abdelfattah NS, Sadda SR; TREX-AMD Study Group. Neovascular age-related macular degeneration management in the third year: final results from the TREX-AMD randomised trial. Br J Ophthalmol. 2018 Apr;102(4):460-464. doi: 10.1136/bjophthalmol-2017-310822. Epub 2017 Aug 4. PMID 28779006

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sixty patients were enrolled between February 2013 and January 2014.
Period: Overall Study
Arm/Group | Monthly IVT Ranibizumab | Treat and Extend IVT Ranibizumab
Started | 20 | 40
Completed | 18 | 28
Not Completed | 2 | 12
Not completed — Adverse Event | 2 | 4
Not completed — Lost to Follow-up | 0 | 3
Not completed — Death | 0 | 3
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Monthly IVT Ranibizumab | Treat and Extend IVT Ranibizumab | Total
Number analyzed (Participants) | 20 | 40 | 60
Age, Continuous [Mean (Full Range); unit: years] | 79 [60 to 96] | 76 [59 to 91] | 77 [59 to 96]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 26 | 38
  Male | 8 | 14 | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Number of Right Eyes Enrolled [Count of Participants; unit: Participants] | 10 | 16 | 26
Number of Participants with Posterior Chamber Intraocular Lenses [Count of Participants; unit: Participants] | 10 | 22 | 32
Diabetes Mellitus [Count of Participants; unit: Participants] | 2 | 9 | 11
Hypertension [Count of Participants; unit: Participants] | 16 | 31 | 47
Early Treatment Diabetic Retinopathy Study Best-Corrected Visual Acuity [Mean (Full Range); unit: letters] | 60.3 [31 to 76] | 59.9 [18 to 78] | 60.0 [18 to 78]
Central Retinal Thickness [Mean (Full Range); unit: microns] | 533 [323 to 839] | 489 [265 to 1007] | 511 [265 to 1007]

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in BCVA by ETDRS Letter Score From Baseline
Description: Mean change in Best-Corrected Visual Acuity (BCVA) by Early Treatment Diabetic Retinopathy Study (ETDRS) letter score from baseline through weeks 24-28, baseline through weeks 48-56, baseline through weeks 72-82, baseline to week 104, baseline through weeks 128-132 and baseline to week 156. The ETDRS protocol is a widely accepted international standard for macular laser photocoagulation treatment. A higher score represents better functioning. The scale ranges from 0 to 100 letters
Time Frame: 6, 12, 18, 24, 30, and 36 months
Population: All participants were included in analysis. Due to participant attrition, missed visits, and variable follow-up intervals in the Treat and Extend arm, the population analyzed at each time point is equal to or smaller than the population still enrolled at that time point.
Measure: Mean (Standard Error); unit: ETDRS BCVA Letters
Arm/Group | Monthly IVT Ranibizumab | Treat and Extend IVT Ranibizumab
Number analyzed (Participants) | 20 | 40
ETDRS BCVA Letters
  Month 6: number analyzed (Participants) | 20 | 36
  Month 6 | 10.5 (1.3) | 7.3 (1.9)
  Month 12: number analyzed (Participants) | 20 | 28
  Month 12 | 9.2 (1.4) | 10.5 (2.0)
  Month 18: number analyzed (Participants) | 18 | 25
  Month 18 | 10.4 (1.9) | 9.0 (3.2)
  Month 24: number analyzed (Participants) | 19 | 23
  Month 24 | 10.5 (1.9) | 8.7 (3.6)
  Month 30: number analyzed (Participants) | 19 | 20
  Month 30 | 9.7 (2.3) | .95 (4.4)
  Month 36: number analyzed (Participants) | 18 | 20
  Month 36 | 8.6 (2.8) | 4.1 (4.0)

2. Secondary Outcome: Incidence and Severity of Adverse Events (Ocular and Non-ocular)
Description: Incidence and severity of adverse events both ocular and non-ocular
Time Frame: 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | Monthly IVT Ranibizumab | Treat and Extend IVT Ranibizumab
Number analyzed (Participants) | 20 | 40
Participants
  Participants Experiencing Serious Ocular AE | 2 | 6
  Participants Experiencing Serious Systemic AE | 7 | 20

3. Secondary Outcome: Total Number of Intravitreal Injections Required
Description: Total number of intravitreal injections required from baseline through weeks 48-57 (week closest to week 52), baseline through week 104 and baseline through week 156.
Time Frame: 12, 24, and 36 months
Population: as for outcome 1
Measure: Mean (Full Range); unit: injections
Arm/Group | Monthly IVT Ranibizumab | Treat and Extend IVT Ranibizumab
Number analyzed (Participants) | 20 | 40
injections
  Month 12: number analyzed (Participants) | 20 | 37
  Month 12 | 13.0 [13 to 13] | 10.1 [7 to 13]
  Month 24: number analyzed (Participants) | 20 | 30
  Month 24 | 25.5 [22 to 27] | 18.6 [10 to 25]
  Month 36: number analyzed (Participants) | 18 | 28
  Month 36 | 31.5 [25 to 39] | 25 [10 to 37]

4. Secondary Outcome: Total Number of Office Visits and Imaging Studies Performed During Study Period
Description: Total number of office visits and imaging studies performed from baseline through weeks 24-28 (week closest to week 26), baseline through weeks 48-56 (week closest to week 52), baseline through weeks 72-82 (week closest to week 78), baseline through week 104, baseline through weeks 128-132 (week closest to week 132) and baseline through week 156
Time Frame: 6, 12, 18, 24, 30, and 36 months
Population: Per protocol, imaging was conducted at each study visit and is assumed to be perfectly correlated with the number of visits. Therefore, only visits were specifically analyzed. Additionally, given the high correlation between number of visits and injections administered (reported previously), this analysis was performed only at M12, M24, and M36.
Measure: Number; unit: scheduled visits completed
Arm/Group | Monthly IVT Ranibizumab | Treat and Extend IVT Ranibizumab
Number analyzed (Participants) | 20 | 40
scheduled visits completed
  Number of Visits through Month 12 | 262 | 364
  Number of Visits through Month 24 | 560 | 838
  Number of Visits through Month 36 | 801 | 1143

5. Secondary Outcome: Percentage of Subjects With Persistent Active Exudation on SD-OCT
Description: Percentage of subjects with persistent active exudation on SD-OCT from baseline through weeks 48-57 (week closest to week 52), baseline through week 104 and baseline through week 156.
Time Frame: 12, 24, and 36 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Monthly IVT Ranibizumab | Treat and Extend IVT Ranibizumab
Number analyzed (Participants) | 20 | 40
Participants
  Month 12: number analyzed (Participants) | 20 | 36
  Month 12 | 3 | 9
  Month 24: number analyzed (Participants) | 19 | 28
  Month 24 | 5 | 9
  Month 36: number analyzed (Participants) | 18 | 28
  Month 36 | 9 | 8

6. Secondary Outcome: Mean Change in Central Foveal Thickness
Description: Mean change in central foveal thickness by SD-OCT from baseline to weeks 48-57, baseline to week 104 and baseline to week 156.
Time Frame: 12, 24, and 36 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: microns
Arm/Group | Monthly IVT Ranibizumab | Treat and Extend IVT Ranibizumab
Number analyzed (Participants) | 20 | 40
microns
  Month 12: number analyzed (Participants) | 19 | 28
  Month 12 | -246 (43) | -173 (31)
  Month 24: number analyzed (Participants) | 18 | 23
  Month 24 | -170 (37) | -170 (37)
  Month 36: number analyzed (Participants) | 18 | 28
  Month 36 | -188 (42) | -183 (32)

7. Secondary Outcome: Percentage of Patients With Persistent Leakage on Fluorescein Angiography
Description: Percentage of subjects with persistent leakage on fluorescein angiography from baseline through weeks 24-28, baseline to weeks 48-56, baseline to weeks 72-82, baseline to week 104, baseline to weeks 128- 132 and baseline to week 156.
Time Frame: 6, 12, 18, 24, 30, and 36 months
Population: This analysis was never performed because we were logistically unable to collect the data.
Arm/Group | Monthly IVT Ranibizumab | Treat and Extend IVT Ranibizumab
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: CNVM Lesion Size
Description: CNVM lesion size at baseline, compared to baseline to weeks 24-28, baseline to weeks 48-56, baseline to weeks 72-82, baseline to week 104, baseline to weeks 128-132 and baseline to week 156, as determined by fluorescein angiography.
Time Frame: 6, 12, 18, 24, 30, and 36 months
Population: This analysis was never performed because we were logistically unable to collect the data.
Arm/Group | Monthly IVT Ranibizumab | Treat and Extend IVT Ranibizumab
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 years (entire study period)
Description: Adverse events were assessed at every study visit during the 3-year study
Arm/Group | Monthly IVT Ranibizumab | Treat and Extend IVT Ranibizumab
All-Cause Mortality (participants affected / at risk) | 0/20 | 3/40
Serious Adverse Events (participants affected / at risk) | 7/20 | 23/40
Other Adverse Events (participants affected / at risk) | 2/20 | 4/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Monthly IVT Ranibizumab (N=20) | Treat and Extend IVT Ranibizumab (N=40)
Unexplained vision loss, left eye (Eye disorders) | 0 (0) | 1 (1)
Temporal arteritis (Vascular disorders) | 0 (0) | 1 (1)
Worsening of gout, cellulitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Retinal pigment epithelium tear (Eye disorders) | 0 (0) | 1 (1)
Severe pneumonia, dehydration, anemia, COPD, emphysema, lung cancer (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchitis and Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Leukocytosis (General disorders) | 1 (1) | 0 (0)
Broken ribs (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Worsening of arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 1 (1)
Abdominal pain (General disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Acute cholecystitis with abnormal liver function tests (Hepatobiliary disorders) | 0 (0) | 1 (1)
Acute varicella zoster encephalitis (Infections and infestations) | 0 (0) | 1 (1)
Worsening of COPD (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Meningitis, urinary tract infection, and congestive heart failure (Infections and infestations) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
(Death) High cervical vertebral fracture w/ severed spinal cord tear in descending aorta (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
(Death) Hemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Subretinal hemorrhage (Eye disorders) | 0 (0) | 1 (1)
(Death) hypoxemia; gastrointestinal bleed; duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Motor vehicle accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Influenza B (Infections and infestations) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Monthly IVT Ranibizumab (N=20) | Treat and Extend IVT Ranibizumab (N=40)
Subretinal hemorrhage (Eye disorders) | 1 (1) | 1 (1)
Progressive macular atrophy (Eye disorders) | 0 (0) | 3 (3)
Hollenhorst plaque (Eye disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The key limitation is the small population analyzed through 3 complete years; subject attrition due to elderly population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2015-01-16): https://cdn.clinicaltrials.gov/large-docs/92/NCT01748292/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2014-10-22): https://cdn.clinicaltrials.gov/large-docs/92/NCT01748292/Prot_SAP_001.pdf